CLINICAL TRIAL: NCT02990013
Title: Comparison of Antimicrobial Activity of AvenovaTM as a Sterile Skin Preparation in Humans
Brief Title: AvenovaTM as a Sterile Skin Preparation Agent
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wendy Lee, Associate Professor of Clinical Ophthalmology & Dermatology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20160881
Record Dates: First submitted 2016-11-29; First posted 2016-12-12 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Cleaning Product Causing Toxic Effect
MeSH Terms: interventions — Povidone-Iodine; Solutions; Chlorhexidine; 2-Propanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment arm (Experimental): All patients will be in the treatment arm where they will be subject to skin testing with various cleansing agents: AvenovaTM , povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol
  Interventions: Device: Avenova; Drug: Povidone-iodine 5% solution; Drug: 4% chlorhexidine; Drug: Isopropyl alcohol

INTERVENTIONS:
Device: Avenova — Subjects will all undergo the treatment arm where their skin will be cleansed with four different agents: AvenovaTM , povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol
  Other Names: hypochlorous acid
Drug: Povidone-iodine 5% solution — Subjects will all undergo the treatment arm where their skin will be cleansed with four different agents: AvenovaTM , povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol
  Other Names: Betadine
Drug: 4% chlorhexidine — Subjects will all undergo the treatment arm where their skin will be cleansed with four different agents: AvenovaTM , povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol
  Other Names: No other names
Drug: Isopropyl alcohol — Subjects will all undergo the treatment arm where their skin will be cleansed with four different agents: AvenovaTM , povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol
  Other Names: No other names

SUMMARY:
Aim 1: To determine in vivo capability of AvenovaTM against common cutaneous microbial biome on human skin

Aim 2: To compare to povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol against AvenovaTM as a sterile skin agent

DETAILED DESCRIPTION:
A total of approximately 30 eligible participants will be identified with clinically-acquired information by Dr. Wendy Lee, an oculoplastic surgeon and aesthetic treatment specialist at Bascom Palmer Eye Institute, during regular clinic visits.

Part One: Patients will have their skin swabbed and then cultured for various skin flora agents. The petri dish will then be swabbed with Avenova to see what percent of skin flora microbe is killed.

Part Two: Patients will have their skin divided into 4 quadrants. The area will be pre-swabbed to monitor microbe growth. Each of 4 quadrants will be cleansed for one minute with AvenovaTM , povidone-iodine 5% solution, 4% chlorhexidine and isopropyl alcohol, then swabbed to monitor for microbe growth.

The swabs will be placed in thioglycollate broth to monitor for bacterial growth. If growth if observed in the thioglycollate, the samples will be cultured on blood agar plates and the bacterial specie(s) identified.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above able to provide informed consent to participate Adults attending Dr. Wendy Lee Oculoplastics Clinic

Exclusion Criteria:

* Adults unable to consent
* Individuals who less than 18 years of age
* Prisoners
* Pregnant women - while these cleansing agents are used on pregnant women as standard cleansing agents, effects to fetus unknown
* Patients currently using oral or topical antimicrobial agents
* History of skin infection to facial injectable of surgery
* Inability to tolerate cleansing procedure
* Inability to sit comfortably for 15 - 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of Avenova to other standard of care cleansing agents: growth vs. no growth | 12 months
  Growth or no growth of bacteria in the thioglycollate broth will be noted for the control and each quadrant after cleansing with the 4 agents listed above.

SECONDARY OUTCOMES:
Bacterial Identification | 12 months
  Positive thioglycollate samples will be cultured on blood agar plates and the bacterial species then identified.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lee, Principal Investigator — Bascom Palmer Eye Institute University of Miami, Miller School of Medicine
Locations (1):
- University of Miami Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Requests can be e-mailed to Dr. Wendy Lee: WLee@med.miami.edu

REFERENCES:
- [Background] Collins LK, Knackstedt TJ, Samie FH. Antiseptic use in Mohs and reconstructive surgery: an American College of Mohs Surgery member survey. Dermatol Surg. 2015 Jan;41(1):164-6. doi: 10.1097/DSS.0000000000000202. No abstract available. PMID 25521104
- [Background] Steinsapir KD, Woodward JA. Chlorhexidine Keratitis: Safety of Chlorhexidine as a Facial Antiseptic. Dermatol Surg. 2017 Jan;43(1):1-6. doi: 10.1097/DSS.0000000000000822. PMID 27399954
- [Background] Kim HJ, Lee JG, Kang JW, Cho HJ, Kim HS, Byeon HK, Yoon JH. Effects of a low concentration hypochlorous Acid nasal irrigation solution on bacteria, fungi, and virus. Laryngoscope. 2008 Oct;118(10):1862-7. doi: 10.1097/MLG.0b013e31817f4d34. PMID 18677274
- [Background] Robson MC, Payne WG, Ko F, Mentis M, Donati G, Shafii SM, Culverhouse S, Wang L, Khosrovi B, Najafi R, Cooper DM, Bassiri M. Hypochlorous Acid as a Potential Wound Care Agent: Part II. Stabilized Hypochlorous Acid: Its Role in Decreasing Tissue Bacterial Bioburden and Overcoming the Inhibition of Infection on Wound Healing. J Burns Wounds. 2007 Apr 11;6:e6. PMID 17492051
- [Background] Debabov D, Noorbakhsh C, Wang L, et al. Avenova™ with Neutrox™ (pure 0.01% HOCl) compared with OTC product (0.02% HOCl). NovaBay Pharmaceuticals, Inc., Emeryville, California, USA.